CLINICAL TRIAL: NCT02448342
Title: Sensible Medical Innovations (Noninvasive) Lung fLuid Status Monitor Allows rEducing Readmission Rate of Heart Failure Patients- a Randomized Controlled Study
Brief Title: Sensible Medical Innovations Lung fLuid Status Monitor Allows rEducing Readmission Rate of Heart Failure Patients
Acronym: SMILE™
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Sensible Medical Innovations Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CL-00100-P
Record Dates: First submitted 2015-05-10; First posted 2015-05-19 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-08

CONDITIONS: Heart Failure
Keywords: Heart Failure; Remote Patient Monitoring; Non Invasive Lung Fluid Status Monitor
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ReDS Guided Treatment (Experimental): After discharge from hospital, patient will perform daily ReDS measurement. Data is automatically transmitted to the secured web portal. Treating physician will follow up on patients' measurements through a secured dedicated web site. Notification messages will be automatically sent by the system to the physician if certain thresholds are crossed (thresholds are physician adjustable). Medications will be adjusted according to defined guidelines. During the study a service center will monitor and support patient adherence and investigators attending to patients' notifications.
  Interventions: Device: Remote Dielectric Sensing (ReDS) Wearable System
- Standard of Care- Control arm (Active Comparator): After discharge from hospital, patient will be followed up and medically managed according to standard of care guidelines.
  Interventions: Device: Remote Dielectric Sensing (ReDS) Wearable System

INTERVENTIONS:
Device: Remote Dielectric Sensing (ReDS) Wearable System — The ReDS device provides noninvasive measurement of lung fluid content. It comprises a wearable vest with embedded sensors and a bedside console, with touch-screen display. A measurement reading is provided within 90sec. Results are shared with the treating physician via a secured web portal.
  Other Names: ReDS; Wearable Vest

SUMMARY:
Multi center, randomized controlled study, to determine if a significant decrease in the rate of heart failure re-hospitalizations occurs during a follow-up period when - ReDS guided treatment is used as an adjunct to standard of care.

DETAILED DESCRIPTION:
The study is designed as a prospective, randomized, controlled, multi-center trial. Patients will be enrolled during an index hospitalization for Acutely decompensated Heart Failure (ADHF) and will be followed for a minimum of 3 months or a maximum of 9 months (until the last patient has completed the 3- month follow-up). Patients will be blinded to ReDS readings values.

Recruitment will take place either during a heart failure hospitalization (see acceptance criteria below) or within 10 days after discharge from a qualifying heart failure hospitalization.

The Remote Dielectric Sensing (ReDS) device provides noninvasive measurement of lung fluid content. It comprises a wearable vest with embedded sensors and a bedside console. A measurement reading is provided within 90sec. Results are shared with the treating physician via a secured web portal.

Study objective is to determine if a significant decrease in the rate of heart failure re-hospitalizations occurs during the entire follow-up period when ReDS guided treatment is used as an adjunct to standard of care (SOC).

Patients will be randomized between two groups before hospital discharge to: ReDS with SOC vs. SOC.

Patient that are randomized to the treatment arm will perform daily ReDS measurement at home. Treating physician will follow up on patients' measurements through a secured dedicated web site. Notification messages will be automatically sent by the system to the physician if certain thresholds are crossed (thresholds are physician adjustable). Medications will be adjusted according to defined guidelines.

Patients that are randomized to the control arm will be followed up and medically managed according to standard of care guidelines.

Both arms scheduled clinical visits and phone follow up:

* A follow up phone call, per current treatment guidelines, will be attempted within 2 days of hospital discharge to obtain information regarding medication reconciliation, Heart Failure (HF) symptoms and other HF management issues (e.g., dietary restrictions).
* An outpatient clinic visit will be scheduled after a week of hospital discharge.
* Study follow-up visits at 1 and 3 months. Follow-up will be continued for enrolled subjects at 6 and 9 months until the last subject has pass through the 3-month follow-up window.

  * At each study follow-up visit, patients will undergo complete physical exam, vital signs, collection of readmission and standard blood tests and QOL questionnaire.

ELIGIBILITY:
Main Inclusion Criteria:

1. Patient has signed informed consent and authorization to use and disclose health information.
2. Patient's physical condition enables him to sit up and lay down with minimal assistance.
3. Diagnosis of HF, with preserved or reduced LVEF, was made at least 30 days prior to enrollment.
4. Patients with LVEF <40% must have been treated at least 30 days prior to enrollment with diuretics and beta-blocker (unless intolerant or contra-indicated) and an ACE-inhibitor or ARB (unless intolerant or contra-indicated).
5. Patient is hospitalized for ADHF requiring significant alteration in heart failure treatment (i.e. diuretics or vasoactive drugs) or up to 10 days post-discharge from an ADHF admission.
6. BNP ≥ 350 pg/ml (NT pro BNP > 1400 pg/ml) at enrollment (within 24h) and/or ≥750 pg/ml any time during the hospital stay (NT-pro BNP >3000 pg/ml).

Note that if a patient is enrolled during a clinic visit rather than during a hospitalization, then the BNP from the index admission is referenced.

Main Exclusion Criteria:

1. Patient has had a cardiac transplantation or VAD implantation.
2. CRT implantation within 90 days prior to screening or planned implantation during study duration.
3. Current or past Pulmonary Embolism in the right lung. Notes: (i) Past pulmonary emboli are defined as identified <6 months prior to enrollment. (ii) past or current tiny, microscopic pulmonary emboli do not exclude a patient. (iii) if a ventilation-perfusion (VQ) scan shows that the lungs are clear, then the exclusion criteria is not met.
4. Diagnosis of Severe Pulmonary Hypertension.
5. STEMI and or CABG within 30 days of screening visit. Note: Type 2 MI due to ADHF is not an exclusion.
6. Chronic renal failure with CrCl<25mL/min, as calculated by the Cockcroft-Gault formula.
7. Chronic home IV therapy or cardiac inotropes or diuretics
8. Physical deformity in the thorax area or lesion that may prevent proper vest application or adjustment (Severe scoliosis/ sensitive sternotomy lesion etc.).
9. Illness/ Condition which may be aggravated or cause significant discomfort by the application of the vest (Rib fractures, with or without flail chest, Severe Osteoporosis).
10. Impaired cognitive ability or any other state that may prevent full compliance with the study protocol, according to investigator's assessment.
11. Patient's habitus out of range due to one or more of the following:

    * Height less than 155cm or higher than 195cm (5.1; 6.4 feet respectively).
    * BMI of less than 22 or more than 36. In case of BMI between 36-38, if the measured vest ruler is not >=4, the exclusion criteria is met.
12. Congenital heart malformations or intra-thoracic mass that would affect the right lung anatomy (Dextrocardia, Lung Carcinoma etc.) including pacemaker box on the right side of the chest.
13. Severe COPD, defined as chronic and continuous home use of O2 (O2 dependancy) and/ or oral steroids. Continuous is defined as 24hours a day, every day.
14. Severe disease / conditions with life expectancy <6 months according to investigator's assessment.
15. Patient is enrolled in another interventional study with permission of study manager (observational or registries are not excluded).
16. Patient HF is managed remotely with another monitoring device or program (for example: Pulmonary/ Lt Atrial pressure monitoring, Weight scale, BNP or bioimpedance).
17. Prisoners and ward of the state

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
The rate of recurrent events of HF readmissions | Entire follow-up period (Expected average of 6.5 months)

SECONDARY OUTCOMES:
Time from discharge until the first event of HF readmissions | Time to event (from discharge until the date of first event of HF readmissions, assessed up to 6.5 months)
Proportions of total days lost to hospitalization due to HF events | Entire follow-up period (Expected average of 6.5 months)
Time from discharge until all-cause mortality | time to event (from time of discharge until the date of first event of HF readmissions, assessed up to 6.5 months)

CONTACTS AND LOCATIONS:
Overall Officials: William Abraham, MD, Principal Investigator — Ohio State University; Aharon (Ronnie) Abbo, MD, Study Director — Sensible Medical Innovations Ltd.
Locations (41):
- United States (41):
  - University of Alabama, Birmingham, Alabama
  - Cedars Sinai, Hollywood, California
  - Scripps Memorial Hospital La Jolla, La Jolla, California
  - Scripps Mercy Hospital San Diego, San Diego, California
  - UCSF Medical Center, Parnassus, San Francisco, California
  - Pacific Heart Institute, Santa Monica, California
  - Yale University Medical Center, New Haven, Connecticut
  - MedStar Heart and Vascular Institute, Washington D.C., District of Columbia
  - Washington DC VA Medical Center, Washington D.C., District of Columbia
  - Memorial Regional Hospital, Hollywood, Florida
  - Encore Research Group, Jacksonville, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Northshore University HealthSystem, Evanston, Illinois
  - Advanced Heart Care Group, Fairview Heights, Illinois
  - Edward Heart Hospital, Naperville, Illinois
  - Prairie Heart Institute / St. John's Hospital, Springfield, Illinois
  - St Elizabeth Healthcare, Edgewood, Kentucky
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - St. Louis Heart and Vascular, St Louis, Missouri
  - Bryan Heart, Lincoln, Nebraska
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Hospital, New Hyde Park, New York
  - Mount Sinai Medical Center, New York, New York
  - Weil Cornell Medical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Suma Health Services, Akron, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Dorothy M. Davis Heart & Lung Research Institute at The Ohio State University Wexner Medical Center, Columbus, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Lancaster General Health Hospital, Lancaster, Pennsylvania
  - Drexel University Medical Center, Philadelphia, Pennsylvania
  - VA Pittsburgh Health System, Pittsburgh, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Pinnacle Health Cardiovascular Institute, Wormleysburg, Pennsylvania
  - Centennial Medical Center - Sarah Cannon Research Institute, Nashville, Tennessee
  - Virginia Cardiovascular Specialties, Midlothian, Virginia
  - Henrico Doctors' Hospital, Richmond, Virginia

REFERENCES:
- [Background] Amir O, Rappaport D, Zafrir B, Abraham WT. A novel approach to monitoring pulmonary congestion in heart failure: initial animal and clinical experiences using remote dielectric sensing technology. Congest Heart Fail. 2013 May-Jun;19(3):149-55. doi: 10.1111/chf.12021. Epub 2013 Jan 25. PMID 23350643
- [Background] Amir O, Azzam ZS, Gaspar T, Faranesh-Abboud S, Andria N, Burkhoff D, Abbo A, Abraham WT. Validation of remote dielectric sensing (ReDS) technology for quantification of lung fluid status: Comparison to high resolution chest computed tomography in patients with and without acute heart failure. Int J Cardiol. 2016 Oct 15;221:841-6. doi: 10.1016/j.ijcard.2016.06.323. Epub 2016 Jul 1. PMID 27434357
- [Background] Amir O, Ben-Gal T, Weinstein JM, Schliamser J, Burkhoff D, Abbo A, Abraham WT. Evaluation of remote dielectric sensing (ReDS) technology-guided therapy for decreasing heart failure re-hospitalizations. Int J Cardiol. 2017 Aug 1;240:279-284. doi: 10.1016/j.ijcard.2017.02.120. Epub 2017 Mar 3. PMID 28341372
- See also: Sponsor web site — http://sensible-medical.com/